CLINICAL TRIAL: NCT04973306
Title: Neoadjuvant Immunotherapy Combined With Chemoradiotherapy Versus Neoadjuvant Chemoradiotherapy for Locally Advanced Resectable Esophageal Squamous Cell Carcinoma (cII-III Stage): A Multi-center Prospective Randomized Clinical Trial
Brief Title: Neoadjuvant Immunotherapy Plus CRT Versus Neoadjuvant CRT for Locally Advanced Resectable ESCC
Acronym: iCROSS
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Peking University Cancer Hospital & Institute (Other); Shanghai Chest Hospital (Other); First Affiliated Hospital of Wenzhou Medical University (Other); Tianjin Medical University Cancer Institute and Hospital (Other); Ningbo Medical Center Lihuili Hospital (Other Government); The First People's Hospital of Changzhou (Other); Zhongshan Hospital (Xiamen), Fudan University (Other); Xuhui Central Hospital, Shanghai (Other); Shanghai Minhang Central Hospital (Other); Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other); Zhejiang Cancer Hospital (Other); Sichuan Cancer Hospital and Research Institute (Other); Tongji Hospital (Other); Sun Yat-sen University (Other); Shanghai Fifth People's Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2021-369R
Record Dates: First submitted 2021-06-28; First posted 2021-07-22 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Esophageal Squamous Cell Carcinoma Stage II; Esophageal Squamous Cell Carcinoma Stage III
Keywords: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Neoadjuvant Therapy; tislelizumab; spartalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neoadjuvant chemoradiotherapy combined with anti-PD-1 antibody (Experimental): Neoadjuvant chemoradiotherapy (NCRT) combined with tislelizumab is performed followed by Ivor-Lewis or Mckeown esophagectomy in enrolled patients.
  Interventions: Procedure: Neoadjuvant Chemoradiotherapy; Drug: Tislelizumab; Procedure: Ivor-Lewis or Mckeown Esophagectomy(Mckeown Esophagectomy recommended)
- Neoadjuvant chemoradiotherapy (Active Comparator): Neoadjuvant chemoradiotherapy (NCRT) is performed followed by Ivor-Lewis or Mckeown esophagectomy in enrolled patients.
  Interventions: Procedure: Neoadjuvant Chemoradiotherapy; Procedure: Ivor-Lewis or Mckeown Esophagectomy(Mckeown Esophagectomy recommended)

INTERVENTIONS:
Procedure: Neoadjuvant Chemoradiotherapy — Chemotherapy: carboplatin (AUC 2 mg/mL per min) and paclitaxel (50 mg/m2 of body-surface area) were administered intravenously for five cycles, starting on days 1, 8, 15, 22, and 29. For each cycle, Carboplatin and paclitaxel were administered 30 minutes apart.
  Radiotherapy: A total radiation dose of 41.4 Gy was given in 23 fractions of 1.8 Gy, 5 days per week (Radiotherapy was performed on the 2nd, 3rd, 4th, 5th, and 6th day in each cycle, and only 3 times in the 5th cycle)
Drug: Tislelizumab — Tislelizumab (200mg/time) was administered intravenously on the 1st and 22nd day.
  The intravenous injection lasts about 30 minutes (micropump is recommended, intravenous bolus is prohibited, duration should be not less than 20 minutes and not more than 60 minutes);
  Other Names: anti-PD-1 antibody
  Arms: Neoadjuvant chemoradiotherapy combined with anti-PD-1 antibody
Procedure: Ivor-Lewis or Mckeown Esophagectomy(Mckeown Esophagectomy recommended) — After neoadjuvant therapy, patients in groups receive Ivor-Lewis or Mckeown Esophagectomy (Mckeown Esophagectomy recommended)

SUMMARY:
The purpose of this study was to evaluate the safety, feasibility and outcome of anti-PD-1 antibody (Tislelizumab, BeiGene) combined with neoadjuvant chemoradiotherapy versus neoadjuvant chemoradiotherapy followed by minimally invasive esophagectomy for locally advanced resectable esophageal squamous cell carcinoma (cII-III Stage) patient.

DETAILED DESCRIPTION:
It is a prospective randomized phase II&III clinical trial sponsored by Shanghai Zhongshan Hospital with other twelve hospitals in China participating in. 476 patients with locally advanced resectable esophageal squamous cell carcinoma (cII-III Stage) are recruited and randomly assigned into the neoadjuvant chemoradiotherapy combined with immunotherapy group (nCRT plus anti-PD-1 Group) and the neoadjuvant chemoradiotherapy group (nCRT Group) according to the proportion of 1:1. The safety, efficacy of protocols and prognosis of patients are compared between the two regimens.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically-confirmed esophageal squamous cell carcinoma and whose tissue samples were taken before treatment;
2. Tumors of the esophagus are located in the thoracic cavity;
3. Pre-treatment stage as clinical II-III (AJCC/UICC 8th Edition)
4. Age is between 18 years and 75 years;
5. Eastern Cooperative Oncology Group (ECOG) performance status 0-1, and expected survival time ≥12 months;
6. Adequate cardiac function. All patients should perform ECG, and those with a cardiac history or ECG abnormality should perform echocardiography with the left ventricular ejection fraction > 50 %;
7. Adequate respiratory function with FEV1≥1.2L, FEV1%≥50% and DLCO≥50% shown in pulmonary function tests ;
8. Adequate bone marrow function (White Blood Cells >4x10^9 /L; Neutrophil >2.0×10^9 /L; Hemoglobin > 90 g/L; platelets>100x10^9 /L);
9. Adequate liver function (Total bilirubin <1.5x Upper Level of Normal (ULN); Aspartate transaminase(AST) and Alanine transaminase (ALT) <1.5x ULN);
10. Adequate renal function (Glomerular filtration rate (CCr) >60 ml/min; serum creatinine (SCr) ≤120 µmol/L);
11. The patient has provided written informed consent and is able to understand and comply with the study;

Exclusion Criteria:

Exclusion Criteria associated with Cancer:

1. Patients with histological non-squamous cell carcinoma;
2. Patients with advanced non-operable or metastatic esophageal cancer;
3. Pre-treatment stage as cM+, cN3 or cT4b(non-curatively-resectable verified by the local surgical investigator, AJCC/UICC 8th Edition) or cTis-1a, cT1bN0;
4. Patients with another previous or current malignant disease which is likely to interfere with treatment or the assessment of response in the judgement of the local surgical investigator;
5. Patients who have received or are receiving other chemotherapy, radiotherapy or targeted therapy;

   Other Exclusion Criteria:
6. Patients with autoimmune diseases history;
7. Recently or currently taking Glucocorticoids or Immunosuppressants;
8. Patients who underwent immunotherapy in the past;
9. Allergy to any antibody drugs or allergy to Paclitaxel and Carboplatin.
10. Past or currently suffering from chronic or recurrent autoimmune diseases;
11. Patients with active infection of immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV); HIV seropositivity; HBV DNA or HCV RNA positive;
12. Patients with organ transplantation (including autologous bone marrow transplantation and peripheral stem cell transplantation);
13. Patients with severe systematic intercurrent disease, such as active infection or poorly controlled diabetes; coagulation disorders; hemorrhagic tendency or under treatment of thrombolysis or anticoagulant therapy;
14. Any patient with a significant medical condition which is thought unlikely to tolerate the therapies. Such as cardiac disease (e.g. symptomatic coronary artery disease or myocardial infarction within last 12 months), clinically-significant lung disease, clinically-significant bone marrow, liver, renal function disorder;
15. Pregnant or lactating women and fertile women who will not be using contraception during the trial;
16. Participation in another intervention clinical trial with interference to the chemotherapeutic or chemoradiotherapeutic intervention during this study or during the last 30 days prior to informed consent;
17. Expected lack of compliance with the protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2022-03-02 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Pathological response rate(pCR) | Up to the date of pathological reports obtained since the date of randomization, up to 12 months
  The resected specimen following neo-adjuvant treatment are assessed by using standardized work up of the resection specimen in the pathology department and standardized histological criteria for tumor regression grading. The degree of histomorphologic regression is clarified into four categories as follows: grade 1, no evidence of vital residual tumor cells (pathological complete response); grade 2, less than 10% vital residual tumor cells; grade 3, 10 to 50%; and grade 4, more than 50%.
Overall survival(OS) | Up to the date of death of any causes since the date of randomization, up to 36 months

SECONDARY OUTCOMES:
Treatment related complications | Up to 1 month after surgery since the data of randomization, up to 13 months
  Number and severity of adverse events that are related to treatment of each patients (including adverse events associated with neoadjuvant chemoradiotherapy, immunotherapy(irAE) and surgery), and hospital re-admission. Treatment-related adverse events as assessed by CTCAE v5.0
Progression-free survival(PFS) | Up to the date of disease recurrence since the date of randomization, up to 36 months
  Disease recurrence is defined as locoregional (esophageal bed or anastomotic or regional lymph nodes) or metastatic (supraclavicular lymph nodes or distant organs)
R0 resection rate | Up to the date of pathological reports obtained since the date of randomization, up to 12 months
  No vital tumor is presented at the proximal, distal, or circumferential resection margin, it is considered to be R0 resection. If a vital tumor is shown at 1 mm or less from the proximal, distal, or circumferential resection margin, it is considered to be microscopically positive (R1).
Number and Location of positive lymph nodes | Up to the date of pathological reports obtained since the date of randomization, up to 12 months
  According to pathological reports, record the number and location of positive lymph nodes
Overall Quality of life | Up to the end of follow-up since the data of surgery, up to 36 months
  Overall Quality of life is respectively evaluated at randomization and 1 month, 3 month, 6 month and yearly after surgery among patients by using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire C-30 Scale (EORTC QLQ-C30)
Quality of life in eating and swallowing function | Up to the end of follow-up since the data of surgery, up to 36 months
  Quality of life in eating and swallowing function is respectively evaluated at randomization and 1 month, 3 month, 6 month and yearly after surgery among patients by using the EORTC QLQ-OES18 Scale
Recurrence-free survival (RFS) | Up to the date of disease recurrence since the date of surgery, up to 36 months
  RFS is defined in resected patients who achieved an R0 or R1 resection as the time interval from surgery to the date of first recurrence (local, regional or distant) or death, whichever comes first.
Correlation between genetic profile and tumor response | Up to the end of follow-up since the data of surgery, up to 36 months
  Genetic profile (assessed by whole exome sequencing, T-cell receptor sequencing, RNA sequencing) .illumina HiSeq and Nanostring platforms will be used to evaluate the patient's genetic profile. The tumor response will be evaluated by an experienced thoracic tumor pathologist in our center through Tumor regression grading (TRG) systems.

CONTACTS AND LOCATIONS:
Overall Officials: Lijie Tan, MD, Principal Investigator — Shanghai Zhongshan Hospital
Locations (1):
- Shanghai Zhongshan Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No
According to the regulations on the management of human genetic resources of the People's Republic of China, we will not be able to share Individual Participant Data

REFERENCES:
- [Background] Chen W, Zheng R, Baade PD, Zhang S, Zeng H, Bray F, Jemal A, Yu XQ, He J. Cancer statistics in China, 2015. CA Cancer J Clin. 2016 Mar-Apr;66(2):115-32. doi: 10.3322/caac.21338. Epub 2016 Jan 25. PMID 26808342
- [Background] van Hagen P, Hulshof MC, van Lanschot JJ, Steyerberg EW, van Berge Henegouwen MI, Wijnhoven BP, Richel DJ, Nieuwenhuijzen GA, Hospers GA, Bonenkamp JJ, Cuesta MA, Blaisse RJ, Busch OR, ten Kate FJ, Creemers GJ, Punt CJ, Plukker JT, Verheul HM, Spillenaar Bilgen EJ, van Dekken H, van der Sangen MJ, Rozema T, Biermann K, Beukema JC, Piet AH, van Rij CM, Reinders JG, Tilanus HW, van der Gaast A; CROSS Group. Preoperative chemoradiotherapy for esophageal or junctional cancer. N Engl J Med. 2012 May 31;366(22):2074-84. doi: 10.1056/NEJMoa1112088. PMID 22646630
- [Background] Liu S, Wen J, Yang H, Li Q, Chen Y, Zhu C, Fang W, Yu Z, Mao W, Xiang J, Han Y, Zhao L, Liu H, Hu Y, Liu M, Fu J, Xi M. Recurrence patterns after neoadjuvant chemoradiotherapy compared with surgery alone in oesophageal squamous cell carcinoma: results from the multicenter phase III trial NEOCRTEC5010. Eur J Cancer. 2020 Oct;138:113-121. doi: 10.1016/j.ejca.2020.08.002. Epub 2020 Aug 30. PMID 32877795
- [Background] McDermott DF, Atkins MB. PD-1 as a potential target in cancer therapy. Cancer Med. 2013 Oct;2(5):662-73. doi: 10.1002/cam4.106. Epub 2013 Jul 21. PMID 24403232
- [Background] Doi T, Piha-Paul SA, Jalal SI, Saraf S, Lunceford J, Koshiji M, Bennouna J. Safety and Antitumor Activity of the Anti-Programmed Death-1 Antibody Pembrolizumab in Patients With Advanced Esophageal Carcinoma. J Clin Oncol. 2018 Jan 1;36(1):61-67. doi: 10.1200/JCO.2017.74.9846. Epub 2017 Nov 8. PMID 29116900
- [Background] Yamamoto S, Kato K. Immuno-oncology for esophageal cancer. Future Oncol. 2020 Nov;16(32):2673-2681. doi: 10.2217/fon-2020-0545. Epub 2020 Aug 11. PMID 32777942
- [Background] Huang J, Xu J, Chen Y, Zhuang W, Zhang Y, Chen Z, Chen J, Zhang H, Niu Z, Fan Q, Lin L, Gu K, Liu Y, Ba Y, Miao Z, Jiang X, Zeng M, Chen J, Fu Z, Gan L, Wang J, Zhan X, Liu T, Li Z, Shen L, Shu Y, Zhang T, Yang Q, Zou J; ESCORT Study Group. Camrelizumab versus investigator's choice of chemotherapy as second-line therapy for advanced or metastatic oesophageal squamous cell carcinoma (ESCORT): a multicentre, randomised, open-label, phase 3 study. Lancet Oncol. 2020 Jun;21(6):832-842. doi: 10.1016/S1470-2045(20)30110-8. Epub 2020 May 13. PMID 32416073
- [Background] Liao XY, Liu CY, He JF, Wang LS, Zhang T. Combination of checkpoint inhibitors with radiotherapy in esophageal squamous cell carcinoma treatment: A novel strategy. Oncol Lett. 2019 Nov;18(5):5011-5021. doi: 10.3892/ol.2019.10893. Epub 2019 Sep 19. PMID 31612012
- [Background] Li C, Zhao S, Zheng Y, Han Y, Chen X, Cheng Z, Wu Y, Feng X, Qi W, Chen K, Xiang J, Li J, Lerut T, Li H. Preoperative pembrolizumab combined with chemoradiotherapy for oesophageal squamous cell carcinoma (PALACE-1). Eur J Cancer. 2021 Feb;144:232-241. doi: 10.1016/j.ejca.2020.11.039. Epub 2020 Dec 26. PMID 33373868